CLINICAL TRIAL: NCT06159322
Title: A Study Investigating the Relationship Between the Antipsychotic Response and Non-invasive Proxies of Neurochemistry in Schizophrenia
Brief Title: Characterizing Response to Antipsychotics in Schizophrenia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Royal Ottawa Mental Health Centre (Other)
Collaborators: The Royal's Institute of Mental Health Research (Other)
Responsible Party: Sponsor
Other Study IDs: 2021033
Record Dates: First submitted 2022-04-10; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Antipsychotic treatment response
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Olanzapine; Clozapine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First-line treatment group: This group will consist of 20 patients with schizophrenia or schizoaffective disorder who are primarily prescribed olanzapine. Treatment will be carried out by the physicians within their circle of care, however, we will record their symptoms as they continue treatment.
  Interventions: Drug: Olanzapine
- Treatment-resistant group: This group will consist of 20 patients with schizophrenia or schizoaffective disorder who are primarily prescribed clozapine due to poor treatment response to first-line antipsychotic agents. Treatment will be carried out by the physicians within their circle of care, however, we will record their symptoms as they continue treatment.
  Interventions: Drug: Clozapine

INTERVENTIONS:
Drug: Olanzapine — Antipsychotic medication
  Other Names: Zyprexa
  Groups: First-line treatment group
Drug: Clozapine — Antipsychotic medication
  Other Names: Clozaril
  Groups: Treatment-resistant group

SUMMARY:
The goal of this research project is to develop MRI-based biomarkers to identify patients with schizophrenia who are most likely to benefit from first-line antipsychotic or clozapine treatment. The MRI sequences (NM-MRI, MRS and rsfMRI) will be created by translating the best scientific evidence into a potential clinical product that has the highest chance of being clinically relevant predictor of treatment response. This study has the potential to significantly improve patient outcomes and reduce unnecessary interventions and costs at the Royal's Integrated Schizophrenia Recovery Program.

DETAILED DESCRIPTION:
Currently, we cannot predict who will get better on first-line antipsychotic versus clozapine treatment. Although much evidence shows that dopamine and glutamate function are related to treatment response in schizophrenia, the utility of neuromelanin sensitive MRI (NM-MRI) as a measure of dopamine and magnetic resonance spectroscopy (MRS) as a measure of glutamate & glycine (a co-agonist of glutamate receptors) in predicting response to treatment have never been measured in the same sample. The evidence suggests that the function of these two neurotransmitter systems partially determines the response to antipsychotic medications. Additionally, an emerging type of resting-state functional MRI (rsfMRI), naturalistic movie-watching, has been shown to outperform traditional rsfMRI for functional connectivity-based prediction of behaviour and will be explored in the current study. Given the background information, our hypotheses are:

1.1) First-line antipsychotic users will have higher dopamine turnover resulting in a higher NM-MRI signal in the substantia nigra relative to clozapine users.

1.2) First-line antipsychotic users will have lower glutamate and/or glycine concentration as indicated by the MRS signal in the dorsal anterior cingulate relative to clozapine users.

ELIGIBILITY:
Inclusion Criteria:

* Are voluntary and competent to consent to the study
* Are between the ages of 18-55
* Are English literate
* Have a diagnosis of schizophrenia or schizoaffective disorder
* Are currently taking primarily olanzapine or clozapine

Exclusion Criteria:

* Medication for the treatment of schizophrenia or schizoaffective disorder has changed in the past month
* Have a significant neurologic, neurodevelopmental, cardiovascular, renal, hepatic, hematological, gastrointestinal, pulmonary, or metabolic-endocrine disorder
* Are pregnant or breastfeeding
* Acquire positive urine test result for all drugs of abuse including cannabis
* Have met DSM-5 criteria for substance use disorder other than tobacco in the last 6 months
* Have a history of significant head trauma with loss of consciousness for more than 5 minutes
* Have any contraindication to MRI
* Have any other condition that in the opinion of the investigator(s) could create a hazard to the subject's safety, endanger the study procedures, or interfere with the interpretation of study results

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals with a diagnosis of schizophrenia or schizoaffective disorder
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Neuromelanin-sensitive magnetic resonance imaging (MRI) contrast-to-noise ratio (CNR) | Will be examined cross-sectionally on an as-recruited basis.
  Indexes dopamine function
Glutamate/glycine magnetic resonance sptrectroscopy (MRS) | Will be examined cross-sectionally on an as-recruited basis.
  Indexes glutamate & glycine concentration

CONTACTS AND LOCATIONS:
Overall Officials: Lauri Tuominen, MD, PhD, Principal Investigator — The Royal's Institute of Mental Health Research; Clifford Cassidy, PhD, Principal Investigator — The Royal's Institute of Mental Health Research
Locations (1):
- The Royal's Institute of Mental Health Research, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.